CLINICAL TRIAL: NCT05922501
Title: A Phase II Study of ISABELA: Isatuximab, Belantamab Mafodotin, Pomalidomide, and Dexamethasone in Relapsed and Refractory Multiple Myeloma
Brief Title: Isatuximab, Bela Maf, Pom, and Dex in Relapsed/Refractory Multiple Myeloma
Acronym: ISABELA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Sanofi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Andrew Yee, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-183
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Relapsed Cancer; Refractory Multiple Myeloma; Multiple Myeloma
Keywords: Relapsed/Refractory; Multiple Myeloma; Relapsed and Refractory
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — isatuximab; belantamab mafodotin; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Isatuximab + Belantamab mafodotin + Pomalidomide + Dexamethasone (Experimental): Isatuximab will be given once daily into your vein (by intravenous infusion) over about 30-60 minutes. This will occur during cycle 1 (cycle equals 28 days) on days 1, 8, 15, and 22 and cycle 2 and onwards days 1 and 15.
  Belantamab mafodotin will be given once every 8 weeks into your vein (by intravenous infusion) over about 60 minutes after completion of isatuximab infusion.
  Pomalidomide will be taken orally once daily during days 1-21 of each cycle.
  Dexamethasone will be taken orally once daily during days 1, 2, 8, 9, 15, 16, 22, and 23 of each cycle.
  Drug diaries will be provided to participants to document information about taking pomalidomide and dexamethasone.
  Interventions: Drug: Isatuximab; Drug: Belantamab mafodotin; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab — An IgG1-derived monoclonal antibody that targets CD38 proteins, administered intravenously.
  Other Names: SAR650984
Drug: Belantamab mafodotin — An antibody-drug conjugate that is the combination of an antibody targeting BCMA and a drug, administered intravenously.
  Other Names: GSK2857916
Drug: Pomalidomide — An immunomodulatory agent, capsule taken orally.
Drug: Dexamethasone — A glucocorticoid which is a substance that stops inflammation cause by immune system disorders, tablet taken orally.

SUMMARY:
The main goal of this phase II study is to evaluate the overall response rate of isatuximab, belantamab mafodotin, pomalidomide, and dexamethasone in relapsed and refractory multiple myeloma. The study drugs provided for research purposes are isatuximab and belantamab mafodotin.

DETAILED DESCRIPTION:
This is a phase II study of isatuximab, belantamab mafodotin, pomalidomide, and dexamethasone in relapsed and refractory multiple myeloma. Approximately 50 participants will take part in this research study. The primary objective is determining the overall response rate of the treatment. Treatment is until progression, adverse events, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Participant has given voluntary signed written informed consent before performance of any study-related procedure that is not part of normal medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to their future medical care.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (see Appendix A).
* Age ≥ 18 years
* Measurable disease of multiple myeloma as defined by at least one of the following:

  * Serum monoclonal protein ≥ 0.5 g/dL. Patients with IgD disease and lower amounts of monoclonal protein may be permitted to enroll with PI approval
  * ≥ 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Involved serum free light chain ≥ 100 mg/L (10 mg/dL) and abnormal serum free light chain ratio
* Previously treated relapsed and refractory multiple myeloma:
* Patients must have received at least one prior line of therapy;
* Prior therapy must include at least 2 cycles of lenalidomide and at least 2 cycles of a proteasome inhibitor (either in separate regimens or within the same regimen); and
* Disease progression on or within 60 days of completion of last therapy.
* ANC ≥ 1000/μL. G-CSF is not permitted within 14 days of screening. Patients with ANC <1000/µL can be considered for screening on a case-by-case basis with additional monitoring, after discussion with and approval from the PI.
* Platelet count ≥ 75,000/µL. Platelet transfusion is not permitted within 7 days of screening.
* Hemoglobin ≥ 8 g/dL. Red blood cell transfusions are permitted to meet eligibility criteria.
* Calculated creatinine clearance of ≥ 30 mL/min by Modified Diet in Renal Disease (MDRD) formula or Cockcroft-Gault formula
* Spot urine (albumin/creatinine ratios (spot urine) < 500 mg/g or urine dipstick negative/trace.
* Patient has adequate hepatic function, as evidenced by each of the following:
* Serum bilirubin values < 1.5 × ULN. Isolated bilirubin ≥ 1.5 × ULN is acceptable if bilirubin is fractionated and direction bilirubin <35%. Patients with elevated bilirubin due to Gilbert's syndrome may be permitted with PI approval (e.g. total bilirubin <3 mg/dL and normal direct bilirubin); and
* Serum aspartate transaminase (ALT) and/or aspartate transaminase (AST) values < 2.5 × the upper limit of normal (ULN) of the institutional laboratory reference range. Patients with elevated bilirubin due to Gilbert's syndrome may be permitted with PI approval (e.g. total bilirubin <3 mg/dL and normal direct bilirubin).
* Must be able to take acetylsalicylic acid (ASA) daily as prophylactic anticoagulation. Patients intolerant to ASA may use low molecular weight heparin, apixaban, rivaroxaban, or equivalent.
* All study participants must be registered into the mandatory Pomalyst REMS program and be willing and able to comply with the requirements of the Pomalyst REMS program.
* Women of childbearing potential (WOCBP) must adhere to the scheduled pregnancy testing as required in the Pomalyst REMS program and agree to use a highly effective method of contraception during the study for 4 months after the last dose of treatment in the study (see Appendix) and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period). A WOCBP must have a negative highly sensitive serum pregnancy test within 72 hours before the first dose of study intervention and agree to use a highly effective method of contraception during the study and for 4 months after the last dose of belantamab mafodotin. Note: non childbearing potential defined as follows (by other than medical reasons):

  * ≥ 45 years of age and has not had menses for > 1 year
  * Patients who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.
* A man who is sexually active with a WOCBP (even if they have undergone a successful vasectomy) must agree to use a barrier method of birth control e.g. either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository for 6 months after receiving the last dose of study drug.
* Male participants must refrain from donating sperm for 6 months after the last dose of study drug.
* Able to swallow capsules whole (pomalidomide capsules cannot be crushed, dissolved or broken).

Exclusion Criteria:

* Participant must not have had current corneal epithelial disease except mild changes in corneal epithelium.
* Participant must not use contact lenses while participating in this study.
* Participants who have had myeloma therapy or investigational drug within 2 weeks prior to start of treatment or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
* Participants who are receiving any investigational agents.
* Prior therapy with anti-CD38 monoclonal antibody within six months. No other multiple myeloma monoclonal antibody therapy within 30 days of start of study treatment.
* Prior therapy with anti-BCMA therapy.
* Plasmapheresis within seven days prior to start of study treatment.
* Primary refractory disease.
* Concomitant high dose corticosteroids. Low dose corticosteroids (maximum dose prednisone 10 mg/day or equivalent) are permitted if given for disorders other than myeloma, e.g. adrenal insufficiency, rheumatoid arthritis, etc.
* Pregnancy or lactation or planned lactation (breastfeeding).
* Prior history of malignancies, other than MM, unless the patient has completed definitive treatment and has been free of the disease for ≥ 3 years. Patients who are free of disease < 3 years may enroll after discussion with and approval of the PI. Exceptions include the following (i.e. the following are eligible to participate):

  * Basal or squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Ductal carcinoma in situ of the breast
  * Incidental histologic finding of prostate cancer (T1a or T1b) managed with surveillance
* Patients with active plasma cell leukemia at time of screening, POEMS syndrome, or primary AL amyloidosis are excluded from this trial.
* Seropositive for HIV infection
* Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]; see exception below). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened for hepatitis B virus (HBV) DNA levels. Those with positive HBV viral load will be excluded. Exception: subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) and a known history of prior HBV vaccination do not need testing for HBV DNA.
* Seropositive for hepatitis C (except in the setting of a sustained virologic response, defined as aviremia at least 12 weeks after completion of antiviral therapy).
* Peripheral neuropathy ≥ grade 2 despite supportive therapy.
* Hypersensitivity to isatuximab, belantamab mafodotin, pomalidomide, or dexamethasone, such as Stevens-Johnson syndrome. Rash to immunomodulatory drug that can be medically managed is allowed.
* Allogeneic stem cell transplant <12 months prior to initiation of study treatment and who have not discontinued immunosuppressive treatment for at least four weeks prior to initiation of study treatment and who are currently dependent on such treatment. Patients may also not have active graft v. host disease (GVHD).
* Autologous stem cell transplant <6 months prior to start of treatment
* Patient has a history of significant cardiovascular, neurological, endocrine, gastrointestinal, respiratory, or inflammatory illness that could preclude study participation, pose an undue medical hazard, or interfere with the interpretation of the study results, including, but not limited to:

  * Congestive heart failure (New York Heart Association [NYHA] Class 3 or 4)
  * Unstable angina
  * Clinically significant, uncontrolled cardiac arrhythmia such a 2nd degree or 3rd degree atrioventricular block
  * Recent (within the preceding 6 months) myocardial infarction or stroke
  * Uncontrolled hypertension
  * Diabetes mellitus with > 2 episodes of ketoacidosis in the preceding 12 months
  * Chronic obstructive pulmonary disease (COPD) requiring > 2 hospitalizations in the preceding 12 months.
  * Unstable liver or biliary disease
  * Active bacterial, viral, or fungal infection
* Patient has any other medical, psychiatric, or social condition that would preclude participation in the study, pose an undue medical hazard, interfere with the conduct of the study, or interfere with interpretation of the study results.
* Major surgery within 4 weeks prior to C1D1.
* Live or live-attenuated vaccine within 30 days prior to C1D1.
* Toxicity from previous anticancer therapy must resolve to baseline levels or to grade ≤1, except for alopecia and peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 4 weeks
  Evaluated per International Myeloma Working Group Response Criteria

SECONDARY OUTCOMES:
Number of Adverse Events | 4 weeks
  Adverse events will be classified and graded according to the CTCAE v.5.0. Frequencies of adverse events will be summarized on all patients who receive any study drug.
Progression Free Survival (PFS) | The time from start of treatment to disease progression or death from any cause, for up to 10 years. Patients who have not progressed or died are censored at the date last known progression-free.
  PFS is defined as the time from start of treatment to disease progression or death from any cause. Patients who have not progressed or died are censored at the date last known progression-free. This is estimated using the Kaplan-Meier method.
Overall survival (OS) | 4 weeks
  OS is defined as the time from start of treatment to death due to any cause or censored at date last known alive. This is estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Yee, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation